CLINICAL TRIAL: NCT02657447
Title: A Phase 1, Open Label, Randomized Study to Assess Pharmacokinetics, Biodistribution and Radiation Dosimetry of Lutetium (177Lu) Lilotomab Satetraxetan (Betalutin®) Radioimmunotherapy in Patients With Relapsed Non-Hodgkin Lymphoma
Brief Title: Dosimetry Study of Betalutin for Treatment of Relapsed Non-Hodgkin Lymphoma (LYMRIT-37-02)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is no longer relevant
Sponsor: Nordic Nanovector (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2013-003908-39
Record Dates: First submitted 2015-12-22; First posted 2016-01-15 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Radioimmunotherapy; Lu-177; Phase I study; Betalutin; ARC; Antibody Radionuclide Conjugate; HH1; Rituximab; 177Lu-DOTA-HH1; Lymphoma; Lymphoma Non-Hodgkin; Immune System Diseases; Follicular Lymphoma; Marginal Zone Lymphoma; Lymphoplasmacytoid; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histological Type; Small Lymphocytic Lymphoma; Classical Mantle Cell Lymphoma; Lilotomab; Lutetium (177Lu) lilotomab satetraxetan
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; AIDS-Related Complex; Lymphoma; Immune System Diseases; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — tetulomab tetraxetan lu-177; Lutetium; Lutetium-177

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Betalutin with lilotomab dose 1 (Experimental): Betalutin 15 MBq/kg b.w. with lilotomab pre-dosing
  Interventions: Drug: Betalutin with lilotomab dose 1
- Arm 2: Betalutin with lilotomab dose 2 (Experimental): Betalutin 15MBq/kg b.w. with lilotomab pre-dosing
  Interventions: Drug: Betalutin with lilotomab dose 2

INTERVENTIONS:
Drug: Betalutin with lilotomab dose 1 — 15 MBq/kg b.w. Betalutin (lutetium (177Lu) lilotomab satetraxetan) single injection, with lilotomab pre-dosing, dose 1
  Other Names: Betalutin; Lymrit 37-02; lutetium (177Lu) lilotomab satetraxetan; HH1; 177Lu-DOTA-HH1
  Arms: Arm 1: Betalutin with lilotomab dose 1
Drug: Betalutin with lilotomab dose 2 — 15 MBq/kg b.w. Betalutin (lutetium (177Lu) lilotomab satetraxetan) single injection, with lilotomab pre-dosing, dose 2
  Other Names: Betalutin; Lymrit 37-02; lutetium (177Lu) lilotomab satetraxetan; HH1; 177Lu-DOTA-HH1
  Arms: Arm 2: Betalutin with lilotomab dose 2

SUMMARY:
This study is a phase I, open label, randomized study to assess pharmacokinetics, biodistribution and radiation dosimetry of lutetium (177Lu) lilotomab satetraxetan (Betalutin®) radioimmunotherapy in patients with relapsed non-Hodgkin lymphoma. The study will also investigate the safety, toxicity and efficacy of Betalutin and pre-dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed (by WHO classification) relapsed indolent non-Hodgkin B-cell lymphoma of following subtypes: Follicular lymphoma (follicular grade I-IIIA), Marginal zone lymphoma (exclusion of MZL if large lymphocytes > 50%), Small lymphocytic lymphoma, Lymphoplasmacytoid and classical mantle cell lymphoma (no blastoid MCL).
2. Requiring initiation of treatment for the NHL.
3. Relapsed after at least one line of therapy including rituximab combination chemotherapy regimen.
4. Exhausted and/or ineligible for all standard treatment options.
5. Not a candidate for an autologous or allogeneic stem cell transplantation. Patients in progression after successful stem cell collection before before high-dose therapy and autologous stem cell transplantation may be considered for enrolment.
6. Age ≥ 18 years..
7. A pre-study ECOG performance status of 0-2. In selected patients an ECOG score of 3 can be acceptable if it is clearly lymphoma-associated at the discretion of the investigator.
8. Life expectancy should be ≥ 3 months.
9. 9. < 25% tumour cells in bone marrow biopsy prior to lilotomab/Betalutin treatment (biopsy taken from a site not previously irradiated).
10. All patients must have at least one bi-dimensionally measurable lesion (>1.5 cm in its largest dimension by CT scan). Patients without such a target lesion can be accepted on an individual basis if histological organ involvement can be evaluated for response e.g. involvement of the skin or the gastrointestinal tract.
11. Women of childbearing potential must:

    * have a negative serum pregnancy test at screening and before Betalutin injection
    * understand that the study medication is expected to have teratogenic risk
    * agree to use, and be able to comply with, highly effective method of birth control with a Pearl-Index ≤ 1%. Contraception is required without interruption, 4 weeks before starting study drug, throughout study drug therapy and for 12 months after end of study drug therapy, even if she has amenorrhoea.
12. Male subjects must agree to use condoms during intercourse throughout study drug therapy and the following 12 months.
13. Patients previously treated with native rituximab are eligible.
14. The patient is willing and able to comply with the protocol, and agrees to return to the hospital for follow-up visits and examination.
15. The patient has been fully informed about the study and has signed the informed consent form.
16. Negative HAMA test.
17. CD37 positive, re-biopsy or test on existing tumour material if not known

Exclusion Criteria:

1. Medical contraindications, including uncontrolled infection, severe cardiac, pulmonary, neurologic, psychiatric or metabolic disease, steroid requiring asthma/allergy, known HIV positive.
2. Laboratory values during screening :

   * Absolute Neutrophil Counts (ANC) ≤ 1.5 x 109 /l
   * Platelet count ≤ 150 x 109 /l
   * Total bilirubin ≥ 30 mmol/l
   * ALP and ALAT ≥ 4x normal level
   * GFR < 60 ml/min/1.73 m2 as measured by the CKD-EPI method.
3. Known or suspected CNS involvement of lymphoma
4. Previous total body irradiation, or irradiation of > 25% of the patient's bone marrow.
5. Chemotherapy, immunotherapy or another investigational drug received within the last 4 weeks prior to the patient entering screening.
6. Earlier treatment with radioimmunotherapy.
7. Exposure to another CD37 targeting drug.
8. Concurrent participation in another therapeutic treatment trial.
9. Previous hematopoietic stem cell transplantation (autologous and allogenic).
10. Pregnant or lactating women.
11. Transformed or potentially transformed NHL from indolent to aggressive
12. Receipt of live, attenuated vaccine within 30 days prior to enrolment
13. Test positive for hepatitis B (HBsAg and anti-HBc)
14. A known hypersensitivity to rituximab, HH1, Betalutin or murine proteins or any excipient used in rituximab, HH1 or Betalutin
15. Malignant disease, other than that being treated in this study. Exceptions include: malignancies that were treated curatively and have not recurred within 3 years prior to study entry; completely resected basal cell and squamous cell skin cancers; completely resected carcinoma in situ of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Dosimetry | 3 weeks
  Estimation of individual tumour/organ uptake and retention of radioactivity.

SECONDARY OUTCOMES:
The number of participants with adverse events as assessed by NCTCAE. | 12 weeks
  Adverse events by treatment group.
Efficacy (Best overall response rate) | 3 months - 1 year
  Best overall response rate by treatment group as measured by Cheson Criteria.
Lilotomab pharmacokinetics | 3 weeks
  Estimation using decay correction measurements

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Buck, Prof. MD, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Universitätsklinikum Würzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahle J, Repetto-Llamazares AH, Mollatt CS, Melhus KB, Bruland OS, Kolstad A, Larsen RH. Evaluating antigen targeting and anti-tumor activity of a new anti-CD37 radioimmunoconjugate against non-Hodgkin's lymphoma. Anticancer Res. 2013 Jan;33(1):85-95. PMID 23267131
- [Background] Repetto-Llamazares AH, Larsen RH, Mollatt C, Lassmann M, Dahle J. Biodistribution and dosimetry of (177)Lu-tetulomab, a new radioimmunoconjugate for treatment of non-Hodgkin lymphoma. Curr Radiopharm. 2013 Mar;6(1):20-7. doi: 10.2174/1874471011306010004. PMID 23256748